CLINICAL TRIAL: NCT06852677
Title: The Effect of Deep Squat and Cross-Legged Sitting on Range of Motion, Pain, and Visceral Functions in Participants With Low Back Pain: A Randomized Experimental Study
Brief Title: Deep Squat, Cross-Legged Sitting and Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ladislav Batalik (Other)
Responsible Party: Sponsor-Investigator, Ladislav Batalik, Principal Investigator, Brno University Hospital
Organization: Brno University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FT-2025-SQUAT-AH
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain; Hip Pain Chronic
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deep Squat (Experimental): Participants in this experimental group will perform deep squat position daily (20 minutes, 6 days per week) for 6 weeks.
  Interventions: Other: Deep Squat position
- Cross-Legged Sitting (Experimental): Participants in this experimental group will perform cross legged position daily (20 minutes, 6 days per week) for 6 weeks.
  Interventions: Other: Cross-legged Sitting
- Control (No Intervention): Participants in this control group won't have any intervention.

INTERVENTIONS:
Other: Deep Squat position — Participants assigned to the deep squat group will perform a cumulative total of 20 minutes of deep squatting per day, six days a week, for six weeks. The squatting time can be divided into multiple shorter sessions throughout the day, with a maximum interval of 48 hours between sessions. Participants will be instructed to maintain an upright posture with heels on the ground, feet shoulder-width apart, and knees aligned with toes. They will be encouraged to gradually increase their squat duration and comfort over time.
  Before starting the intervention, participants will receive standardized instructions on proper squat form to ensure safety and maximize benefits. Their compliance will be monitored through a training diary in the experimental (Tulkit) app.
  Arms: Deep Squat
Other: Cross-legged Sitting — Participants assigned to the cross-legged sitting group will perform a cumulative total of 20 minutes of cross-legged sitting per day, six days a week, for six weeks. The squatting time can be divided into multiple shorter sessions throughout the day, with a maximum interval of 48 hours between sessions. Participants will be instructed to maintain an upright posture while sitting. They will be encouraged to gradually increase their cross-legged sitting duration and comfort over time.
  Before starting the intervention, participants will receive standardized instructions on proper sitting form to ensure safety and maximize benefits. Their compliance will be monitored through a training diary in the experimental (Tulkit) app.
  Arms: Cross-Legged Sitting

SUMMARY:
The goal of this randomized experimental study is to learn if regular deep squat or cross-legged sitting practice can improve mobility, reduce pain, and enhance visceral functions in adults with chronic low back pain (LBP). The main questions it aims to answer are:

Does practicing deep squat or cross-legged sitting increase joint mobility (hip, spine, ankle) and flexibility? Does it reduce pain levels in the lumbar spine and hip region? Does it improve visceral functions related to digestion and bowel movements? Researchers will compare a deep squat group, a cross-legged sitting group, and a control group to see if these interventions lead to significant improvements in mobility, pain reduction, and visceral function compared to no intervention.

Participants will:

Be randomly assigned to one of three groups (deep squat, cross-legged sitting, or control).

Practice their assigned position for 20 minutes per day, 6 days a week, for 6 weeks.

Undergo baseline and post-intervention assessments, including mobility tests, pain evaluation, and quality-of-life questionnaires.

DETAILED DESCRIPTION:
This randomized experimental study explores the effects of deep squat and cross-legged sitting practice on musculoskeletal mobility, pain perception, and visceral functions in adults with chronic low back pain (LBP). By examining these interventions over a six-week period, the study seeks to determine their potential role as non-pharmacological strategies for managing chronic pain and mobility limitations.

Participants will receive structured guidance to ensure proper execution of the assigned positions and adherence to the intervention protocol. Standardized assessments will be conducted before and after the intervention to evaluate changes in joint mobility, flexibility, pain levels, and quality of life.

The study is designed to contribute to evidence-based rehabilitation practices, offering insights into how simple, posture-based exercises might improve physical function and well-being. Findings may have implications for physiotherapy, rehabilitation, and self-management strategies in individuals with chronic LBP.

ELIGIBILITY:
Inclusion Criteria:

* age 20-60 years, chronic lower back or hip pain lasting at least 3 months, presence of bowel problems at least twice a month for at least 3 months)

Exclusion Criteria:

* acute health problem, pregnancy, hip or knee TEP, patellofemoral syndrome or recent lower limb surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for Pain (VAS) | Change from baseline to 6 weeks
  A scale for measuring the intensity or frequency of pain.
WBLT (The Weight-bearing lunge test) | Change from baseline to 6 weeks
  The Weight-bearing lunge test (WBLT) is used to assess the dorsiflexion range of movement at the ankle joint.
36-Item Short Form Survey (SF-36) | Change from baseline to 6 weeks
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures.
The Patient Assessment of Constipation Quality of Life (PAC-QOL) questionnaire | Change from baseline to 6 weeks
  PAC-QOL is the most validated and the most specific tool for measuring the quality of life of patients with constipation.

SECONDARY OUTCOMES:
Goniometry | Change from baseline to 6 weeks
  Measuring the range of movement (ROM) in hip joints.
Sitting-rising test | Change from baseline to 6 weeks
  Clinical test which provides a significant and efficient prediction of mortality risk in the elderly. It measure the ability to sit and rise up with minimum support.
Sit and reach test | Change from baseline to 6 weeks
  The sit and reach test measures flexibility by having a person sit with their legs straight and reaching forward as far as possible. The distance reached is recorded to assess flexibility, with longer reaches indicating greater flexibility.
Patrick (FABER) test | Change from baseline to 6 weeks
  Clinical pain provocation test designed to assist in diagnosing of pathologies in the hip, lumbar spine, and sacroiliac joint.
Schober test | Change from baseline to 6 weeks
  The Schober test is classically used to determine if there is a decrease in lumbar spine range of motion (flexion).
Stibor test | Change from baseline to 6 weeks
  The Stibor test is classically used to determine if there is a decrease in lumbar and thoracic spine range of motion (flexion).

CONTACTS AND LOCATIONS:
Overall Officials: Adéla Haňurová, BSc., Study Director — LF MUNI
Locations (1):
- University hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No